CLINICAL TRIAL: NCT05914922
Title: Musculoskeletal (MSK) Educational Tool and Impact on Patients Randomized Control Trial - Pilot Study
Brief Title: Wadey RCT MSK Short Case Simulations With FMED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Veronica Wadey, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5777
Record Dates: First submitted 2023-05-05; First posted 2023-06-22 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Musculoskeletal Diseases or Conditions
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Phase I pertained to the development of authentic MSK case presentations. These cases were formulated into case presentations and a full content review was completed for each of the 20 MSK conditions. Phase II will now assess the impact of the case simulations on learning and patient care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMRL CTL-PGY1 (Post Graduate Year 1) and FMRL CTL - PGY2 (Post Graduate Year 2) (No Intervention): This arm of participants reflects family medicine resident learners (FMRLs) who will not be exposed to the 1-20 MSK case simulations.
- FMRL EXP - PGY1 and FMRL EXP - PGY2 (Experimental): This arm of participants reflects family medicine resident learners (FMRLs) who will be exposed to the 1-20 MSK case simulations.
  Interventions: Other: Educational Tool

INTERVENTIONS:
Other: Educational Tool — 20 MSK short case simulations were developed based on authentic patient experiences. Strategies to optimize learning of MSK conditions to prepare learners for real-world clinical encounters would be important for family medicine resident learners. To address this need, 20 case simulations of 15 minute duration were developed. This study will determine if an online educational tool may be impactful for determining competency of family medicine resident learners in developing skills and knowledge of 20 MSK conditions while also determining if the tool impacts patient care and satisfaction.
  Arms: FMRL EXP - PGY1 and FMRL EXP - PGY2

SUMMARY:
Study Agent/ Intervention/ Procedure The educational tool consisted of 20 short (MSK) case simulations of 15 minutes duration reflecting conditions of the upper extremity; lower extremity; spine; trauma and MSK infections were developed, reviewed and integrated into links that also contained demographic questionnaires; pre and post simulation knowledge questions and learner satisfaction surveys.

Outcome Measures

1. Demographic questionnaire for the Learner;
2. 100 MCQ (multiple-choice questionnaire) reflecting the same questions contained in the 20 MSK Short Case Simulations
3. Pre/Post multiple choice question knowledge questionnaire
4. Learner satisfaction questionnaire
5. Patient experience and satisfaction questionnaire - QR Code
6. Educator evaluation questionnaire - QR Code
7. Focus group questionnaire

Primary Objectives

1. To determine if learners working through the 20 MSK Short Case Simulations delivered through on-line links would improve their knowledge, skills and satisfaction in learning how to identify and initially manage patients with various MSK conditions when compared to learners not exposed to the same educational tool.
2. To determine patients' experience undergoing one of the 20 MSK assessments and initial management of their various MSK conditions by the learners and their satisfaction in receiving their initial care management in both groups
3. To determine if the assessment and initial management of the 20 MSK conditions by the learners on the patients was deemed to be competent by the educators in both groups

DETAILED DESCRIPTION:
This study is an educational study and the intervention is the 20 Short Case Simulations. The educational tool consists of 20 short (MSK) case simulations of 15 minutes duration reflecting conditions of the upper extremity; lower extremity; spine; trauma and MSK infections. They've been developed, reviewed and integrated into links that also contain demographic questionnaires; pre and post simulation knowledge questions and learner satisfaction surveys. MSK complaints comprise up to 30% to 40% of primary care visits. Despite this, MSK curriculum vary widely among institutions, and there is little consistency in how physicians in training are prepared to treat MSK disorders. To address this need, these modules were developed specifically for frontline healthcare providers and a full content review was completed to generate an educational tool. The review and refinement process indicated the presence of a statistical difference when comparing post to pre-test knowledge scores; high internal consistency (Chronbach Alpha) and strong satisfaction scores among all participant learners.

Primary Hypothesis:

1. The study hypotheses that the family medicine resident learners being exposed at the start of an academic year to the MSK short case simulations will benefit their assessment and initial management of patients with 20 MSK conditions and that patient experiences will be enhanced when compared to family resident learners not exposed to the same educational tool.

Secondary Hypotheses:

1. The study hypothesize that the confounding variable of self-initiated learning of MSK content by family medicine residents not exposed to the 20 MSK case simulations may result in an increase in knowledge and skills and patient satisfaction.
2. The study further hypothesize that self-directed learning on the part of both CTL (Control) and EXP (Experimental) groups may lead to increase in knowledge and skills that may be a confounding variable reflected in the retention T3 scores.

The study is a Randomized Control Trial. Learners from the SBHSC Family Medicine Residency Training Program (FMRLs) will be recruited into this educational study from July 2nd, 2023 through to May 2024. Patients undergoing assessment and initial management of one of the 20 MSK Short Case Simulations will be recruited during the same study time period of June 2023 through to March 1 2024. Educators providing supervision of the FMRLs (Family Medicine Residents) and management of patients' MSK conditions will be recruited to participate during the same time period of July 2, 2023 through to March 1, 2024. Study Agent/ Intervention/ Procedure The educational tool consisted of 20 short (MSK) case simulations of 15 minutes duration reflecting conditions of the upper extremity; lower extremity; spine; trauma and MSK infections were developed, reviewed and integrated into links that also contained demographic questionnaires; pre and post simulation knowledge questions and learner satisfaction surveys.

Outcome Measures

1. Demographic questionnaire for the Learner;
2. 100 MCQ questionnaire reflecting the same questions contained in the 20 MSK Short Case Simulations
3. Pre/Post multiple choice question knowledge questionnaire
4. Learner satisfaction questionnaire
5. Patient experience and satisfaction questionnaire - QR Code
6. Educator evaluation questionnaire - QR Code
7. Focus group questionnaire

Sample Size Calculation:

N=24 Data Analysis

* Survey Monkey will be used to collect and analyze the data and SAS ( Statistical Analysis System) Version 9.4 or later will be used for statistical analyses
* QR Code will be utilized to collect the information from the patients in the learning environments where MSK conditions are being assessed and initially managed
* QR codes will be provided to the education supervisors after each clinical encounter of the FMRL to be assessed for competence
* Qualitative analysis will be done assessing for knowledge and skills resulting from the MSK Short Case Simulations
* Qualitative analysis will be completed on the focus group data that will determine information pertaining to the overall learning experience

ELIGIBILITY:
Inclusion Criteria:

* Patients with an MSK condition included in the education tool of MSK Short Case Simulations 1-20 (Upper extremity; lower extremity; axial skeleton; trauma and MSK infections Patients) seen either in a family medicine clinic; emergency department; clinical ward in the hospital setting or sporting event at which FMRL were covering from a learners perspective
* Patients assessed by FMRLs between the months of July 2023 through to March 2024
* Patient must be free of cognitive impairment and be able to complete an English survey or have a translator present to assist with the translation
* Electronic devices to accommodate QR codes

Exclusion Criteria:

* non-English speaking participants
* an inability to complete QR codes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-02 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Participant demographics | up to 7 months
  Questionnaire (Qualitative analyses)
Pre and Post-test questionnaires for each of the 20 MSK short case simulations - paired T-tests | up to 7 months
  Knowledge questions
Satisfaction questionnaire for EXP group on the educational experience of the MSK case simulations- qualitative analyses | up to 7 months
  The participants completing the 20 MSK short case simulations will complete a satisfaction questionnaire of the case simulations
Patient experience of their individual clinical encounter with the FMRL | up to 7 months
  the patients will complete a link to a QR code (5 minutes) and indicate their level of satisfaction of their clinical encounter with the FMRL
Educator evaluation of a FMRL | up to 7 months
  An educator who would normally supervisor the FMRL with patients would complete a link to a QR code (2 minutes) and indicate the competency of the FMRL
Focus group | up to 7 months
  All participants will meet at the end of the study/academic year to review the process and their participation in the study

CONTACTS AND LOCATIONS:
Overall Officials: Veronica M Wadey, MD,MA, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu V, Goto K, Carek S, Petrizzi M, Deck JW, Sulapas I, DeStefano S, DeCastro AO, Rooks BJ, Mainous AG 3rd, Kulshreshtha A. Family Medicine Musculoskeletal Medicine Education: A CERA Study. Fam Med. 2022 May;54(5):369-375. doi: 10.22454/FamMed.2022.975755. PMID 35536622
- [Background] Sabesan VJ, Schrotenboer A, Habeck J, Lombardo D, Stine S, Jildeh TR, Meiyappan A. Musculoskeletal Education in Medical Schools: A Survey of Allopathic and Osteopathic Medical Students. J Am Acad Orthop Surg Glob Res Rev. 2018 Jun 28;2(6):e019. doi: 10.5435/JAAOSGlobal-D-18-00019. eCollection 2018 Jun. PMID 30211396
- [Background] De Inocencio J. Epidemiology of musculoskeletal pain in primary care. Arch Dis Child. 2004 May;89(5):431-4. doi: 10.1136/adc.2003.028860. PMID 15102634
- [Background] Matheny JM, Brinker MR, Elliott MN, Blake R, Rowane MP. Confidence of graduating family practice residents in their management of musculoskeletal conditions. Am J Orthop (Belle Mead NJ). 2000 Dec;29(12):945-52. PMID 11140349
- [Background] Glazier RH, Dalby DM, Badley EM, Hawker GA, Bell MJ, Buchbinder R. Determinants of physician confidence in the primary care management of musculoskeletal disorders. J Rheumatol. 1996 Feb;23(2):351-6. PMID 8882045
- [Background] Freedman KB, Bernstein J. Educational deficiencies in musculoskeletal medicine. J Bone Joint Surg Am. 2002 Apr;84(4):604-8. doi: 10.2106/00004623-200204000-00015. PMID 11940622
- [Background] Watts SA, Zhang Z. Competency in musculoskeletal and sports medicine: evaluating a PGY-1 curriculum. Fam Med. 2011 Oct;43(9):659-63. PMID 22002779
- [Background] Day CS, Yeh AC. Evidence of educational inadequacies in region-specific musculoskeletal medicine. Clin Orthop Relat Res. 2008 Oct;466(10):2542-7. doi: 10.1007/s11999-008-0379-0. Epub 2008 Jul 18. PMID 18636305
- [Background] Connolly N, Abdalla ME. Impact of COVID-19 on medical education in different income countries: a scoping review of the literature. Med Educ Online. 2022 Dec;27(1):2040192. doi: 10.1080/10872981.2022.2040192. PMID 35317712
- [Background] Wadey VM, Tang ET, Abelseth G, Dev P, Olshen RA, Walker D. Canadian multidisciplinary core curriculum for musculoskeletal health. J Rheumatol. 2007 Mar;34(3):567-80. Epub 2006 Dec 15. PMID 17183615
- [Background] Rules of Thumb, Gerald van Belle, 2002, Wiley
- [Background] Visit-Specific Satisfaction Instrument (VSQ-9) | RAND